CLINICAL TRIAL: NCT06435117
Title: Cancer Prevention Among Individuals with Mental Ill-health: Co-adapting and Implementing Patient Navigation for Primary Cancer Prevention
Brief Title: Cancer Prevention Among Individuals with Mental Ill-health: Patient Navigation for Primary Cancer Prevention
Acronym: CO-CAPTAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Collaborators: Senior Europa Sociedad Limitada (Unknown); Prolepsis Institute for Preventive, Environmental and Occupational Medicine (Other); Universitat Politècnica de València (Other); STICHTING INTERNATIONAL FOUNDATION FOR INTEGRATED CARE (Unknown); Medical University of Lodz (Other); Consejería de Familia, Juventud y Política Social, Comunidad de Madrid (Unknown); Servicio Madrileño de Salud, Madrid, Spain (Other); Fundacion para la Investigacion e Innovacion Biosanitaria de Atencion Primaria (Unknown); Mental Health Europe - Sante Mentale Europe (Unknown); University Mental Health Research Institute, Athens, Greece (Other); Fundacion para el Fomento en Asturias de la Investigacion Cientifica Aplicada y Tecnologia (Unknown); Consejeria de Salud - Principado de Asturias (Unknown); Servicio de Salud del Principado de Asturias (Unknown)
Responsible Party: Principal Investigator, Igor Grabovac, Project coordinator, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 101104784
Record Dates: First submitted 2024-03-28; First posted 2024-05-30 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-05

CONDITIONS: Cancer
Keywords: Europe; Prevention; Cancer; Cancer prevention; Primary prevention; Mental health; Mental health problems; Patient Navigation; Implementation science; Co-design; Longitudinal; Person-centered
MeSH Terms: conditions — Neoplasms; Psychological Well-Being | interventions — Patient Navigation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- People with mental ill-health (Other): All people with mental ill-health aged 18 or older who visit one of the recruitment sites will be asked to participate. Further participants will be recruited through partner organizations (non-governmental organisations, patient groups and professional organisations) involved in care for individuals with mental ill-health, as well as personal contacts. Additionally, healthcare professionals involved in care of people with mental ill-health will be asked to participate in the qualitative part of the study.
  Interventions: Other: Patient Navigation

INTERVENTIONS:
Other: Patient Navigation — CO-CAPTAIN focuses on co-designing and piloting and evaluating the implementation of patient navigation (PN) for primary cancer prevention in people with mental ill-health. Patient Navigators, trained professionals with experience working with people with mental ill-health, will assist people with mental ill-health in gaining access to and utilizing appropriate primary cancer prevention measures offered within the respective healthcare and social system (including smoking cessation and physical activity and nutritional interventions). For this purpose, Patient Navigators will offer regular appointment with participants, apply motivational interviewing and aid in accessing appropriate materials while aiming at empowering participants in taking an active role and making better and more informed decisions regarding their health.

SUMMARY:
Prevention is essential for reducing cancer-related mortality. However, people with mental ill-health often face difficulties in accessing cancer prevention services. The EU-funded CO-CAPTAIN project aims to co-adapt and implement the Patient Navigation Model for primary cancer prevention in this underserved population. This evidence-based and patient-centred intervention aims to support patient empowerment through removal of systemic barriers, provide social support and promote timely access to primary prevention services.

DETAILED DESCRIPTION:
Cancer and mental ill-health constitute leading public health problems in Europe. More than 84 million people in the European Union (EU) report living with an on-going mental ill-health condition. While issues concerning mental health are of great importance, they often overshadow physical problems that people with mental ill-health face. Such is cancer, which is more prevalent in people with mental ill-health and is also the second most common cause of death in this population. People with mental ill-health often have difficulties in accessing quality cancer prevention services, but are also additionally overlooked in research which makes them overall an underserved population. What data is available, shows that potential reasons for these higher cancer morbidity and mortality rates are linked to more engagement in risky health behaviour (especially higher prevalence of smoking as well as overweight and obesity) but also experiences of significant barriers when accessing the highly fragmented heath care systems.

Timely and evidence-based preventive strategies including optimizing health care pathways provide a solution to the high cancer morbidity and could improve overall health outcomes in this disadvantaged population. One such mixed-skill strategy is Patient Navigation. Therefore, the overall goal of the CO-CAPTAIN project is to co-adapt the Patient Navigation (PN) model focusing on primary cancer prevention and to see if this model can prove to be beneficial in supporting individuals with mental ill-health through care services to reduce cancer risk factors by increasing knowledge, health literacy and empowerment. The Patient Navigation Model is an innovative, evidence-based and patient-centred intervention, which supports patient empowerment through removal of systemic barriers, providing social support and promoting timely access to primary prevention services. Based on implementation science and utilizing the Consolidated Framework for Implementation (CFIR) as well as the Reach, Effectiveness, Adoption, Implementation and Maintenance (RE-AIM) frameworks, the CO-CAPTAIN project aims to reduce the gap in health inequalities for people with mental ill-health by reducing cancer burden and improving overall health, which will, in turn, reduce associated costs across health and social care systems in Europe. Moreover, the CO-CAPTAIN project aims to harness the transformative potential of the integrated care pathways in cancer as well as provide health and social care policy recommendations for the adoption and implementation of the Patient Navigation Model across Europe.

The adapted Patient Navigation Model will be implemented in four European countries (Austria, Greece, Poland, Spain) and its potential to enable and improve access and utilization of primary cancer prevention measures for people with mental ill-health will be evaluated. The study will employ a mixed-methods design allowing for both exploratory and confirmatory research.

The project has been funded by the HORIZON EUROPE Framework Program (Call: Research and Innovation actions supporting the implementation of the Mission on Cancer (HORIZON-MISS-2022-CANCER-01-01) - Improving and upscaling primary prevention of cancer through implementation research) and is coordinated by the Medical University of Vienna.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Individuals who have been diagnosed with one or more mental disorders OR healthcare professionals involved in care of individuals with mental ill-health
* Sufficient knowledge of language

Exclusion Criteria:

* Individuals unable to give consent due to diminished capacity
* Individuals who do not provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1240 (Estimated)
Dates: Start 2024-06-24 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Health data of participants as assessed by self-report or electronic health reports | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in health outcomes and socio-economic risk factors in the course of study participation. Next to socio-demographic data, participants will indicate their health status, alcohol consumption, sexual risk behavior, sun exposure, and vaccination status by self-report or electronic health reports.
Nutritional intake of participants as assessed by the Rapid Prime Diet Quality Score Screener (rPDQS) | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in the health outcome nutritional intake. Nutritional intake will be assessed by the Rapid Prime Diet Quality Score Screener (rPDQS; range: 0-52, where higher values indicate healthier nutritional intake).
Smoking behavior of participants as assessed by the Fagerström Test for Nicotine Dependence (FND) | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in the health outcome smoking behavior. Smoking behavior will be assessed by the Fagerström Test for Nicotine Dependence (FND; range: 0-10, where higher values indicate higher nicotine dependence).
Physical activity of participants as assessed by the International Physical Activity Questionnaire (IPAQ) | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in the health outcome physical activity. Physical activity will be assessed by the International Physical Activity Questionnaire (IPAQ; range: 0-19278 MET minutes per week, where higher values indicate more time spent on physical activity).
Depressive symptoms of participants as assessed by the Patient Health Questionnaire (PHQ-9) | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in the health outcome depressive symptoms. Depressive symptoms will be assessed by the Patient Health Questionnaire (PHQ-9; range: 0-27, where a higher score indicates more severe depressive symptoms).
Generalized anxiety of participants as assessed by the 7-item anxiety scale (GAD-7) | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in the health outcome generalized anxiety. Generalized anxiety will be assessed by the 7-item anxiety scale (GAD-7; range: 0-21, where higher values indicate more severe anxiety symptoms).
Health-related anxiety of participants as assessed by the Whiteley Index (Whiteley-6-R) | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in the health outcome health-related anxiety. Health-related anxiety will be assessed by items from the Whiteley Index (Whiteley-6-R; range: 0-24, where higher values indicate more health anxiety symptoms).
(Health-related) Quality of life of participants as assessed by the World Health Organization Quality of Life Brief Version (WHO-QOL-BREF) | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in (health-related) quality of life. (Health-related) Quality of life will be assessed by items from the World Health Organization Quality of Life Brief Version (WHO-QOL-BREF; range: 4-20, where higher values indicate higher quality of life).
(Health-related) Quality of life of participants as assessed by the descriptive system of the EuroQol - 5 Dimensions - 5 Levels (EQ-5D-5L) | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in (health-related) quality of life. (Health-related) Quality of life will be assessed by items from the descriptive system of the EuroQol - 5 Dimensions - 5 Levels (EQ-5D-5L, where each dimension has a range from 1-5, where a higher value indicates more severe problems).
(Health-related) Quality of life of participants as assessed by the EQ visual analogue scale of the EuroQol - 5 Dimensions - 5 Levels (EQ-5D-5L) | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in (health-related) quality of life. (Health-related) Quality of life will be assessed by items from the EQ visual analogue scale of the EuroQol - 5 Dimensions - 5 Levels (EQ-5D-5L, range: 0-100, where higher values indicate better subjective health).
Self-efficacy of participants as assessed by the General Self-Efficacy Scale (GSES) | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in self-efficacy. Self-efficacy will be assessed by items from the General Self-Efficacy Scale (GSES; range: 10-40, where higher values indicate higher perceived self-efficacy).
Feeling understood and supported by healthcare providers as part of health literacy of participants as assessed by the Feeling understood and supported by healthcare providers (HPS) scale of the Health Literacy Questionnaire (HLQ) | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in feeling understood and supported by healthcare providers (HPS) as part of health literacy. HPS as part of health literacy will be assessed by items of the HPS scale from the Health Literacy Questionnaire (HLQ, range of the mean score: 1-4, where higher values indicate higher perceived HPS).
Having sufficient information to manage one's own health as part of health literacy of participants as assessed by the Having sufficient information to manage my health (HSI) scale of the Health Literacy Questionnaire (HLQ) | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in having sufficient information to manage one's own health as part of health literacy. Having sufficient information to manage my health (HSI) as part of health literacy will be assessed by items of the HSI scale from the Health Literacy Questionnaire (HLQ, range of the mean score: 1-4, where higher values indicate higher perceived HSI).
Actively managing one's own health as part of health literacy of participants as assessed by the Actively managing my health (AMH) scale of the Health Literacy Questionnaire (HLQ) | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in actively managing one's own health as part of health literacy. Actively managing my health (AMH) as part of health literacy will be assessed by items of the AMH scale from the Health Literacy Questionnaire (HLQ, range of the mean score: 1-4, where higher values indicate higher perceived AMH).
Social support as part of health literacy of participants as assessed by the Social support of health scale of the Health Literacy Questionnaire (HLQ) | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in social support as part of health literacy. Social support as part of health literacy will be assessed by items of the social support of health scale from the Health Literacy Questionnaire (HLQ, range of the mean score: 1-4, where higher values indicate higher perceived social support for health).
Appraisal of health information as part of health literacy of participants as assessed by the Appraisal of health information (CA) scale of the Health Literacy Questionnaire (HLQ) | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in appraisal of health information as part of health literacy. Appraisal of health information (CA) as part of health literacy will be assessed by items of the CA scale from the Health Literacy Questionnaire (HLQ, range of the mean score: 1-4, where higher values indicate higher perceived CA).
Ability to actively engage with healthcare providers as part of health literacy of participants as assessed by the Ability to actively engage with healthcare providers (AE) scale of the Health Literacy Questionnaire (HLQ) | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in the ability to actively engage with healthcare providers as part of health literacy. Ability to actively engage with healthcare providers (AE) as part of health literacy will be assessed by items of the AE scale from the Health Literacy Questionnaire (HLQ, range of the mean score: 1-5, where higher values indicate higher perceived AE).
Navigating the healthcare system as part of health literacy of participants as assessed by the Navigating the healthcare system (NHS) scale of the Health Literacy Questionnaire (HLQ) | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in the ability to navigate the healthcare system as part of health literacy. Navigating the healthcare system (NHS) as part of health literacy will be assessed by items of the NHS scale from the Health Literacy Questionnaire (HLQ, range of the mean score: 1-5, where higher values indicate higher perceived NHS).
Ability to find good health information as part of health literacy of participants as assessed by the Ability to find good health information (FHI) scale of the Health Literacy Questionnaire (HLQ) | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in the ability to find good health information as part of health literacy. Ability to find good health information (FHI) as part of health literacy will be assessed by items of the FHI scale from the Health Literacy Questionnaire (HLQ, range of the mean score: 1-5, where higher values indicate higher perceived FHI).
Understand health information well enough to know what to do as part of health literacy of participants as assessed by the Understand health information well enough to know what to do (UHI) scale of the Health Literacy Questionnaire (HLQ) | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in the ability to understand health information well enough to know what to do as part of health literacy. Understanding health information well enough to know what to do as part of health literacy will be assessed by items of the Understand health information well enough to know what to do (UHI) scale from the Health Literacy Questionnaire (HLQ, range of the mean score: 1-5, where higher values indicate higher perceived UHI).
Use of healthcare services of participants as assessed by self-reports | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in use of healthcare services. Use of healthcare services will be assessed by self-reports.
Cost-effectiveness and cost-utility of the Patient Navigation Model for primary cancer prevention in people with mental ill-health as assessed by an economic evaluation | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by evaluating cost-effectiveness and cost-utility. To assess cost-effectiveness and cost-utility of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, an economic evaluation will be carried out by analyzing health outcomes and costs (healthcare costs, cancer costs, burden).
Satisfaction with care of participants as assessed by self-reports and items from the Patient Satisfaction Questionnaire Short Form (PSQ-18) | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in satisfaction with care. Satisfaction with care will be assessed by self-reports and items from the Patient Satisfaction Questionnaire Short Form (PSQ-18, range of the mean score: 1-5, where higher scores indicate higher satisfaction with medical care).
Discrimination experiences of participants as assessed by self-reports | 18 months
  To evaluate the clinical utility/effectiveness of the Patient Navigation Model for primary cancer prevention in people with mental ill-health, the extent to which people with mental ill-health benefitted from the intervention will be assessed by investigating changes in discrimination experiences. Discrimination experiences will be assessed by self-reports.
Facilitators of the Patient Navigation Model as experienced by participants and assessed by qualitative semi-structured interviews | 18 months
  The co-adapted Patient Navigation Model will be evaluated by assessing facilitators of the intervention to determine its effectiveness. Experiences of people with mental ill-health, navigators, and healthcare professionals involved in care of people with mental ill-health will be considered. Qualitative data will be gathered using semi-structured interviews.
Barriers of the Patient Navigation Model as experienced by participants and assessed by qualitative semi-structured interviews | 18 months
  The co-adapted Patient Navigation Model will be evaluated by assessing barriers of the intervention to determine its effectiveness. Experiences of people with mental ill-health, navigators, and healthcare professionals involved in care of people with mental ill-health will be considered. Qualitative data will be gathered using semi-structured interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Igor Grabovac, MD, PhD, Principal Investigator — Medical University of Vienna
Locations (9):
- Austria (3):
  - Hietzing Hospital, Vienna
  - LOGIN - Verein zur Gesundheitsförderung und sozialen Integration, Vienna
  - Medical University of Vienna, Vienna
- Greece (3):
  - Mental Health Clinic, Athens
  - The Day Hospital, Athens
  - The Guest House / Protected apartments, Athens
- The Association of Youth and People with Mental Problems, Their Families and Friends POMOST, Lodz, Poland
- Spain (2):
  - General Directorate of Social Services, council of family, youth and social affairs, community of Madrid (DGSSI-CM), Madrid
  - Servicio Madrileño de Salud (SERMAS), Madrid

IPD SHARING:
Plan to Share IPD: Yes
Upon request from other researchers, the principal investigator may provide study materials and data in an anonymised and limited form, while adhering to the Data Security Department of the Medical University of Vienna.
Supporting Information: Study Protocol, ICF
Time Frame: Accessibility is expected after completion of the study as well as of related publications. Only data that does not allow identification of participants will be made available.
Access Criteria: Upon request

REFERENCES:
- See also: HORIZON EUROPE — https://cordis.europa.eu/project/id/101104784